CLINICAL TRIAL: NCT02648178
Title: Evaluation of Appeal and Impact of E-Cigarettes Among Chronic Smokers With Smoking-Related Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, James D. Sargent, Professor of Pediatric Oncology, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D15154
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Nicotine Dependence, Other Tobacco Product; Bladder Cancer; Lung Cancer; Cancer of Head and Neck
MeSH Terms: conditions — Tobacco Use Disorder; Urinary Bladder Neoplasms; Lung Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HALO G6 (Active Comparator): HALO cigalike model
  Interventions: Device: HALO
- HALO Triton (Active Comparator): HALO tank model
  Interventions: Device: HALO

INTERVENTIONS:
Device: HALO — HALO manufactures e-cigarettes which will be distributed to patients. Two products, the G6 and tank model will be used.

SUMMARY:
This study will test feasibility, in smokers with lung, head & neck, and bladder cancers, that examines the effect of e-cigarette substitution, on measures of smoking-related toxicity and medical outcomes. The aim of the study is to determine the appeal of e-cigarettes compared to regular combustible cigarettes.

DETAILED DESCRIPTION:
The aim of the study is to determine the appeal of e-cigarettes compared to combustible cigarettes as measured by the degree to which patients succeed in reducing their cigarette consumption over the 9 weeks they are supplied with product, along with their consumption of e-cigarettes. We will measure past use of e-cigarettes and cigarettes at baseline, 3, 6, 9, and 12 weeks. We will also assess the effect of e-cigarette substitution on toxicity by measuring expired carbon monoxide and urine NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol) , a carcinogenic metabolite of cigarette smoke.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of lung, head & neck, or bladder cancer within the past 5 years.
2. AJCC (American Joint Committee on Cancer) stages I-IV
3. Daily Smoking (at least 10 cigarettes per day for 10 years) and breath CO (carbon monoxide) greater than or equal to 9 ppm
4. Does not wish to quit smoking now (anyone wishing to quit smoking will be referred for smoking cessation counselling through the DHMC (Dartmouth Hitchcock Medical Center) program)
5. May be receiving anti-cancer agents
6. Age 18 or older
7. Fluent in English;
8. Patient must be capable and willing to provide informed written consent for study participation;
9. Able to participate in study visits

Exclusion Criteria:

1. Cancer surgery planned in the next 9 weeks;
2. Treatment with radiation planned for the next 9 weeks,
3. Actively trying to quit smoking, or planning to in the next 30 days. (If a subject reports that they plan to quit smoking in the next 30 days, we will call them after the 30 days to see if they are still trying to quit.)
4. Any use of e-cigarettes in the past 30 days,
5. Pregnant or trying to get pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Sargent, MD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ecigarette Use: Enrolled participants using the e-cigarette.
Period: Overall Study
Arm/Group | Ecigarette Use
Started | 19
Completed | 10
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Ecigarette Use
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Cigarette Smoking Given 10 or More E-cigarette Sessions in a Day
Description: Participants report of daily cigarette and e-cigarette use for the previous 7 days at each study time-point (baseline and 3, 6, 9, and 12 weeks post-baseline) will be averaged to create usual daily cigarette. Mixed-effects linear regression with a random effect at the participant level will be used to assess the association between usual cigarette use (dependent variable) and usually e-cigarette use (independent predictor) over the study period while accounting for the repeated measures within subject. The model will be fit using restricted maximum likelihood. Time will be included in the model as continuous and categorical, separately, and we assess for stability of the association between cigarette use and e-cigarette over time by including an interaction term between e-cigarette use and time in the model.
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: number of Daily Cigarettes
Arm/Group | Ecigarette Use
Number analyzed (Participants) | 13
number of Daily Cigarettes | 4.37 [3.58 to 5.16]
Statistical Analysis 1: Comparison: Ecigarette Use; Test type: Other — We used a linear mixed model to estimate associations between cigarette smoking and that of e-cigarette smoking, by week and their interactions. We also used the same model to estimate association between biomarkers such as NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol), Nicotine, Cotinine, Hydro and Creatinine and CO (Carbon Monoxide) level,by week and their interactions; We tested whether there were significant associations between cigarette smoking and e-cigarette smoking, as well as whether there were significant associations between biomarkers mentioned above with CO level; We provided estimated values of coefficients from model and their 95% confidence intervals; We used a linear mixed model to estimate associations between cigarette smoking and that of e-cigarette smoking, week and their interactions. We also used the same model to estimate association between biomarkers such as NNAL, Nicotine, Cotinine, Hydro and Creatinine and CO level, week and their interactions

2. Primary Outcome: Average Number of E-cigarettes Used Per Day
Description: Average number of e-cigarettes used per day over the 12 week period
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: ecig sessions per day
Arm/Group | Ecigarette Use
Number analyzed (Participants) | 13
ecig sessions per day | 5.04 [3.13 to 6.94]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Ecigarette Use
All-Cause Mortality (participants affected / at risk) | 1/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecigarette Use (N=19)
Death (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT02648178/Prot_SAP_000.pdf